CLINICAL TRIAL: NCT05550103
Title: Effect of Serial Remote Ischemic Conditioning on Dynamic Cerebral Autoregulation in Patients With Intravenous Thrombolysis (SRICDCA-IVT)
Acronym: SRICDCA-IVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRICDCA-IVT
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): RIC+Standard medical treatment. Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 consecutive days from thrombolysis.
  Interventions: Procedure: Remote ischemic conditioning; Other: Standard medical treatment
- Sham RIC+Standard medical treatment (Placebo Comparator): Sham RIC+Standard medical treatment. Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 consecutive days from thrombolysis.
  Interventions: Procedure: Sham remote ischemic conditioning; Other: Standard medical treatment

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC+Standard medical treatment
Other: Standard medical treatment — Standard medical treatment

SUMMARY:
The purpose of this study is to determine the effect of serial remote ischemic conditioning on dynamic cerebral autoregulation in patients with intravenous thrombolysis with alteplase.

DETAILED DESCRIPTION:
In this study, cases of ischemic stroke who undergo intravenous thrombolysis with alteplase within 4.5 hours from the onset are included according to the principle of random, and parallel control. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 7 consecutive days. Both groups underwent dynamic cerebral autoregulation measurements at days 1,3,and 7 of onset and recorded the relevant indexes. We aimed to determine the effect of serial remote ischemic conditioning on dynamic cerebral autoregulation in patients with intravenous thrombolysis with alteplase.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age≥18 years, regardless of sex;
* 2) Patients with clinically definite diagnosis of acute ischemic stroke and undergo intravenous thrombolysis with alteplase in 4.5 hours;
* 3) Baseline mRs 2-5; and Premorbid mRS ≤ 1；
* 4) Baseline NIHSS>= 4, and <= 24;
* 5) Signed and dated informed consent is obtained;

Exclusion Criteria:

* 1) Patients who have the contraindication of intravenous thrombolysis with alteplase;
* 2) Patients with consciousness disorder or restlessness who cannot cooperate with dynamic cerebral autoregulation;
* 3) Patients whose stable cerebral blood flow velocity envelope cannot be obtained by transcranial Doppler ultrasound or whose cerevral blood vessels have not been detected;
* 4) The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb. Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
* 5) Pregnant or lactating women;
* 6) Previous remote ischemic conditioning therapy or similar treatment;
* 7) Laboratory indicators are not qualified: Alanine transaminase (ALT) or glutamic-oxalacetic transaminase (AST) continued to rise more than 3 times the upper limit of normal, Serum creatinine > 265 umol/l (> 3.0 mg/dl);
* 8) Previous history of atrial fibrillation or ECG showing atrial fibrillation or arrhythmia;
* 9) Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons;
* 10) Unwilling to be followed up or treated for poor compliance;
* 11) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission;
* 12) Other conditions that the researchers think are not suitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Dynamic cerebral autoregulation parameter | 0-7 days
  Dynamic cerebral auto-regulation parameters derived from transfer function analysis. Continuous cerebral blood flow velocities of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Transfer function analysis will be used to derive the autoregulatory parameters.

SECONDARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) | 0-7 days
  National Institute of Health stroke scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.
modified Rankin Scale (mRS) | 0-90 days
  modified Rankin Scale (mRS) ranged from 0 to 6, a low value represents a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China